CLINICAL TRIAL: NCT02053467
Title: Building Capacity for Specialized Services Through eConsultation
Acronym: eConsult
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bruyère Health Research Institute. (Other)
Collaborators: Ontario Ministry of Health and Long Term Care (Other Government); The Ottawa Hospital (Other); Ontario Medical Association (Other); Champlain Local Health Integration Network (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 20130674-01H
Record Dates: First submitted 2014-01-30; First posted 2014-02-03 (Estimated); Last update posted 2019-02-05 (Actual); Status verified 2017-02

CONDITIONS: Health Services Research
Keywords: eConsultation; Specialist care; Primary health care; Reducing wait times for specialist care; Reducing referral rates

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- eConsult (Experimental): Physicians randomized to the intervention will have access to the Champlain BASE eConsult service right away (pending completion of an orientation session)
  Interventions: Other: Champlain BASE eConsult Service
- Control (No Intervention): Physicians randomized to the control group will use their standard referral practices for one year after randomization and only then will be given the option to use eConsult.

INTERVENTIONS:
Other: Champlain BASE eConsult Service — After undergoing registration, which includes orientation and brief training on the use of the service, physicians randomized to intervention arm will be able to submit patient-specific clinical questions to specialists through a secure, web-based application. Specialists are asked to respond within 7 days and, for each eConsult, are able to: (1) provide a recommendation, (2) request more information, or (3) recommend a face-to-face referral. The communication between PCPs and specialists is iterative and the discussion can occur back and forth until, ultimately, the PCP closes the case.
  Other Names: A secure Microsoft SharePoint network
  Arms: eConsult

SUMMARY:
The consultation-referral process is complex, involving several steps including 1) the PCP recognizing the need for specialist advice/intervention, 2) patient agreement on seeing the specialist, 3) referral letter and information sent to specialist, 4) appointment booked and communicated, 5) patient visit(s) with the specialist and 6) communication back to the PCP.

There are many factors during this process which limit the effectiveness and efficiency of patient care. These include inequitable access for patients and providers, long wait times before specialist advice received/implemented, delayed communication and mismatched consult expectations. These gaps result in significant breakdowns in transitions of care, inappropriate treatment, patient dissatisfaction and potential harm. Moreover, not all individuals are willing or able to travel to see specialists in a large academic medical centre even when recommended by the PCP.

Electronic consultation (eConsult) service is a form of asynchronous communication whereby primary care providers (PCP) and specialists can communicate directly about a patient through a secure web-based application. eConsult has the potential for improving transitions in care through improved communication ensuring that patients are seen by the right specialist, when necessary, with the right information and in a timely manner. The goal of this project is to evaluate the impact of eConsult on specialist referral rates using health administrative data.

DETAILED DESCRIPTION:
Research Question: What is the impact of an electronic consultation (eConsult) service on referral rates from primary care doctors to specialists?

The objective of this study is to assess the impact of eConsult service on referral rates using a randomized controlled trial (RCT) of eConsult versus usual referral practices. We hypothesized that access to eConsult would lead to a decrease in referral requests for face-to-face specialist visits from primary care providers in the intervention group.

Trial Design: This study is a parallel arm RCT that recruited family physicians in Ontario to use the Champlain BASE™ eConsult service. Physicians will be randomized 1:1 to either the intervention or control arm between January 31, 2014 and September 26, 2014. Although originally intended as a stepped wedge RCT, the design was changed to a parallel arm before and after RCT due to the fact that randomization could not be performed at a discrete time point for all participants.

Intervention: In 2009 our team began developing, implementing, and evaluating an innovative eHealth solution called the Champlain BASE™ (Building Access to Specialists through eConsultation) eConsult service. eConsult is a form of asynchronous communication whereby primary care providers (PCP) and specialists can communicate directly about a patient through a secure web-based application. Specifically, PCPs can submit a patient question (usually for a patient who would otherwise have been referred) to a specialty service via a web-based portal. They can attach any additional information (e.g. photos, test results, Electronic Medical Record-generated letter). The case is assigned to a specialist, who receives an email notification prompting them to access the case via the secure site. Specialists are expected to provide an answer within one week. They can reply to the question, request additional information, or recommend a referral, and advise the PCP on other matters such as medication changes, additional tests, or other critical actions to be completed before the face-to-face specialty care appointment. PCPs ultimately decide how to apply the specialist's suggestion and when the case can be closed. Specialists are compensated on a pro-rated hourly basis. The communication between PCPs and specialists is iterative and the discussion can occur back and forth until, ultimately, the PCP closes the case. After undergoing registration, which included orientation and brief training on the use of the service, physicians randomized to the intervention group will receive access to eConsult right away (pending completion of an orientation session), while those randomized to the control group will use standard referral practices for one year after randomization and then will receive an option to use eConsult in the second year. The intervention period for the treatment group therefore will last one year following the enrollment/randomization period.The pre-randomization period will be 12 months in duration for both groups.

Sample size: With 50 physicians in each arm, assuming an average of 800 patients per physician for a total of 80,000 patients seen, the investigators will achieve 80% power to detect an absolute reduction in referrals of 6 per 100 patients from a control arm referral rate of 31 per 100 patients, estimated from a previous study, using a two-sided significance level of 5% and assuming a between-provider coefficient of variation of 0.38.

Data sources: The following databases from the Institute for Clinical Evaluative Sciences (ICES, ices.on.ca) will be used to obtain physician and patient characteristics: Registered Persons Database, containing demographic data for all residents eligible for provincial health care; Ontario Health Insurance Program (OHIP) billing claims system capturing approximately 95% of physician services in Ontario; the Client Agency Program Enrolment Registry and Corporate Provider Database, for patient enrolment with individual primary care physicians; and the ICES Physician Database, containing physician demographic information, training, and practice setting. 2006 Statistics Canada Census data will be used to assign income quintile to patients based on their postal code. These datasets will be linked using unique encoded identifiers and analyzed at ICES. In addition, the Champlain BASE™ eConsult utilization data, which is routinely collected by the service, will be used to identify the physicians in each group (treatment and control) as well as the date of randomization which was used to identify the relevant 12 month long pre- and post-intervention periods for referral rates assessment.

Data Analysis: All analyses will estimate Intent to Treat (ITT) effects. Descriptive statistics will be generated to describe patient and physician characteristics at the time of randomization for the two groups: eConsult and control. The primary outcome, referral rate per 100 patients seen to all medical specialties available via eConsult service, will be analyzed using a repeated measures multivariable random effects negative binomial regression model. The unit of analysis will be the provider.To account for underlying secular/time trends in the rate of referrals over the study period, the effect of the intervention will be expressed as the between-arm difference in the change in referral rates from the pre- to post-intervention periods (both 12 months in duration).

ELIGIBILITY:
Inclusion Criteria:

* Any practicing primary care provider (PCP) in Ontario who is not currently registered to use the Champlain BASE eConsult service may be recruited to participate in the research study, beginning with the Champlain and South East Local Health Integration Networks.

Exclusion Criteria:

* Those not meeting the inclusion criteria.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2014-01-01; Primary Completion 2016-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Specialist referral rate per 100 patients seen (to medical specialties available through eConsult) | 24 months
  Specialist referral rate defined as the total number of referrals to all medical specialties available through eConsult service during the study period per 100 unique patients (not encounters) seen. The denominator "patients seen" included patients who were seen at least once during the assessment period (baseline or post-intervention).

SECONDARY OUTCOMES:
Specialist referral rates per 100 patients seen (to all medical specialties) | 24 months
  Specialist referral rate defined as the total number of referrals to all medical specialties per 100 unique patients (not encounters) seen. The denominator "patients seen" included patients who were seen at least once during the assessment period (baseline or post-intervention).

CONTACTS AND LOCATIONS:
Overall Officials: Clare Liddy, MD, Principal Investigator — Bruyere Research Institute, C. T. Lamont Primary Health Care Research Centre
Locations (1):
- Bruyere Research Institute, C. T. Lamont Primary Health Care Research Centre, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Liddy C, Maranger J, Afkham A, Keely E. Ten steps to establishing an e-consultation service to improve access to specialist care. Telemed J E Health. 2013 Dec;19(12):982-90. doi: 10.1089/tmj.2013.0056. Epub 2013 Sep 27. PMID 24073898
- [Background] Keely E, Liddy C, Afkham A. Utilization, benefits, and impact of an e-consultation service across diverse specialties and primary care providers. Telemed J E Health. 2013 Oct;19(10):733-8. doi: 10.1089/tmj.2013.0007. Epub 2013 Aug 27. PMID 23980939
- [Background] Liddy C, Rowan MS, Afkham A, Maranger J, Keely E. Building access to specialist care through e-consultation. Open Med. 2013 Jan 8;7(1):e1-8. Print 2013. PMID 23687533
- [Derived] Liddy C, Moroz I, Keely E, Taljaard M, Deri Armstrong C, Afkham A, Kendall CE. Understanding the impact of a multispecialty electronic consultation service on family physician referral rates to specialists: a randomized controlled trial using health administrative data. Trials. 2019 Jun 10;20(1):348. doi: 10.1186/s13063-019-3393-5. PMID 31182123